CLINICAL TRIAL: NCT07137091
Title: Motion for Recovery: The Impact of Gyrokinesis on Childhood Cancer-Related Fatigue.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, Assisstant professor, MTI University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005915
Record Dates: First submitted 2025-08-16; First posted 2025-08-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gyrokinesis exercise (Experimental): Structure of a Gyrokinesis Session
  1. Warm-Up:
     * Begin with gentle seated movements to prepare the body.
     * Focus on awakening the spine with small circles and undulating motions, coordinating with deep breathing.
  2. Seated Exercises:
     * Perform a series of exercises on a stool or chair.
     * Emphasize spinal articulation, pelvic tilts, and side bends while maintaining rhythmic breathing.
  3. Floor Work:
     * Transition to mat-based exercises focusing on core strength and flexibility.
     * Incorporate movements like leg lifts, spirals, and arching motions to engage different muscle groups.
  4. Standing Series:
     * Conclude with standing exercises to enhance balance and full-body integration.
     * Use spiral movements and weight shifts to energize the body and improve posture.
  Interventions: Other: Gyrokinesis exercise
- control group (No Intervention): No intervention

INTERVENTIONS:
Other: Gyrokinesis exercise — 1. Warm-Up:
     * Begin with gentle seated movements to prepare the body.
     * Focus on awakening the spine with small circles and undulating motions, coordinating with deep breathing.
  2. Seated Exercises:
     * Perform a series of exercises on a stool or chair.
     * Emphasize spinal articulation, pelvic tilts, and side bends while maintaining rhythmic breathing.
  3. Floor Work:
     * Transition to mat-based exercises focusing on core strength and flexibility.
     * Incorporate movements like leg lifts, spirals, and arching motions to engage different muscle groups.
  4. Standing Series:
     * Conclude with standing exercises to enhance balance and full-body integration.
     * Use spiral movements and weight shifts to energize the body and improve posture.
  Arms: Gyrokinesis exercise

SUMMARY:
CRF influences engagement in everyday activities, mood, sleep, social relations, school attendance, academic achievement, and quality of life . It was significantly associated with low health-related quality of life in pediatric cancer patients including leukemia . Since attention to managing cRF has been drawn, only a few non-pharmacological strategies were tested for their effectiveness in reducing cRF among children. Physical activity (Pa) has been proven to be the most effective strategy . Yet adherence to Pa remains problematic.

DETAILED DESCRIPTION:
Childhood cancer-related fatigue (CCRF) is a prevalent condition that affects the quality of life in pediatric cancer patients. Gyrokinesis, a holistic exercise method that incorporates principles from yoga, tai chi, and dance, offers potential benefits in managing fatigue through gentle movement and breath work.

According to The American Cancer Society (ACS) provides comprehensive guidelines for cancer training load .The intensity of the exercise refers to the amount of energy expended when performing the activity4. It can be measured subjectively with a self-reported estimate of effort called the rate of perceived exertion on a scale of 1-10. Low-intensity exercise refers to physical activity or effort performed at 1-3 times the intensity of baseline resting energy expenditure (<3 mets-for example, walking). Moderate-intensity exercise refers to physical activity 3-6 times the intensity of baseline, which requires a moderate amount of effort and noticeably accelerates the heart rate (3-6 mets-for example, brisk walking or cycling). Vigorous-intensity exercise refers to physical activity 6 or more times baseline, which requires a large amount of effort and causes rapid breathing and a substantial increase in heart rate (>6 mets-for example, running or jumping rope)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed and treated for a brain tumor during childhood or adolescence (0-≤18 years).
* Treated for a PBT during the previous 10 years, starting from date of diagnosis.

  * Aged ≥6 years 0 months at the start of the trial.
  * Off therapy/active treatment for pediatric brain tumor (PBT) for 12 months at the start of the trial.
  * No known signs of clinical or radiological tumor progression at last follow-up.
  * Danish is the sole or primary language (enabling provision of validated assessment tools).
  * Patient and family have provided consent for inclusion in the trial.

Exclusion Criteria:

* History of recent poorly controlled seizures.
* Motor tics or Tourette syndrome (including family history of tic disorder).

  * Known diagnosis of Attention Deficit/Hyperactivity Disorder or Autism Spectrum Disorder.
  * Known diagnosis of Full Scale Intelligence Quotient (FSIQ) of <50.
  * Pregnancy. Participants known to be pregnant or breastfeeding at screening/registration will not enrolled

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Pediatric quality of life multidimensional fatigue scale (peds QLMFS): | at baseline and at 8 weeks
  CRF was measured using the valid and reliable Arabic version of peds QlMFs . It is an 18-item questionnaire including 'general fatigue', 'sleep/rest fatigue', and 'cognitive fatigue'. The three child self-report versions were used depending on the child's age: 5-7 years (young child), 8-12 years (child), and 13-18 years (adolescent). Higher scores indicate less intense fatigue symptoms . Before the cOViD-19 pandemic, a paper-based appropriate version of the scale was completed by children. During the pandemic, the questionnaires were offered to the participants through a link sent to the parent's phones to eliminate cross-infection.

SECONDARY OUTCOMES:
The six-minute walk test (6-MWT) | at baseline and at 8 weeks
  The 6-MWt is a functional test that measures the functional capacity/endurance and submaximal or maximal effort needed to perform activities of daily living . The primary outcome of this test is the distance covered in meters. a lower score reflects less functional capacity conceptualizing the child's inability to actively participate in functional activities due to cRF .the test is valid and reliable for children with cancer. Two small cones were placed to mark the starting and end points for a 25-meter-long corridor. The heart rate (hR) and oxygen saturation (spO2) were measured 10 min before and one minute after the 6-MWt according to the guidelines of the American thoracic society (ats).
Emotional Well-Being | at baseline and at 8 weeks
  The Children's Depression Inventory (CDI) is scored by summing the responses to its 27 items, with each item having three options scored 0, 1, or 2, resulting in a total score ranging from 0 to 54. Higher scores indicate more severe depressive symptoms.
Blood panel test | at baseline and at 8 weeks
  Blood samples were collected before and after the experiment to assess changes in serotonin and cortisol levels, as described previously . Venous blood samples (6 mL) were obtained from the antecubital vein using a disposable syringe between 8:00 a.m. and 10:00 a.m. after a fasting period of at least 8 hr. Capillary blood samples were also obtained via the fingertip method, with a minimum volume of 0.3 μL collected for analysis using a portable lactate analyzer. Cortisol can also be measured in the blood, with samples typically taken in the morning when levels peak

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy ,Cairo University, Cairo, Egypt